CLINICAL TRIAL: NCT05994430
Title: The Effect of End-of-Life Care Awareness Education on Knowledge, Attitudes, and Behaviors of Intensive Care Nurses: A Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Cansu POLAT DÜNYA, Assisstant of Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20221401
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: End-of-life Care
Keywords: end-of-life; knowledge; attitude; behaviour; intensive care unit nurse; awarnness
MeSH Terms: conditions — Death; Behavior | interventions — Critical Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): The "End-of-Life Care Awareness Training Program in Intensive Care" prepared by the researchers in line with the End-of-Life Nursing Education-Intensive Care (ELNEC-Critical Care) program was applied to the intensive care nurses in the training group. The program was implemented online by determining a common day and time interval suitable for the working hours of the nurses. Half an hour before the training, nurses were reminded of the training topics of the relevant week, time, and Zoom link address via text message.
  40-60 minutes one day a week for 4 weeks in the training program; Week 1: Introduction of the training program and palliative care nursing in intensive care Week 2: Pain management and management of other symptoms (respiratory, gastrointestinal, etc.) Week 3 Communication, cultural and spiritual issues Week 4: Loss, grief, mourning, and ethics were covered.
  Interventions: Other: End-of-life care awareness training in intensive care
- Control Group (No Intervention): Intensive care nurses in the control group did not receive any intervention during the study. The nurses in this group continued to participate in routine in-service trainings. Similar to the training group, the post-test forms/scales "End-of-Life Care Knowledge Test and the Scale of Attitudes and Behaviors of Intensive Care Nurses Towards End-of-Life Care" were administered to the intensive care nurses in the control group in order to determine the changes in the levels of knowledge, attitudes and behaviors towards end-of-life care over time and to compare them with the training group.

INTERVENTIONS:
Other: End-of-life care awareness training in intensive care — End-of-life care awareness training in intensive care
  Arms: Training Group

SUMMARY:
This study was designed as a prospective randomized controlled study in order to evaluate the effect of end-of-life care awareness training to be given to intensive care nurses on the knowledge levels, attitudes, and behaviors of nurses. The study was conducted between May and July 2023 with 76 nurses working in the Anesthesia and Reanimation Intensive Care Unit, General Intensive Care Unit, and Cardiovascular Surgery Intensive Care Unit of Van Training and Research Hospital, who met the inclusion criteria. The hypotheses of this research:

H1: End-of-life care awareness training increases the knowledge level of intensive care nurses about end-of-life care.

H2: End-of-life care awareness training positively affects intensive care nurses' attitudes toward end-of-life care.

H3: End-of-life care awareness training positively affects the behaviors of intensive care nurses towards end-of-life care.

Nurses who completed their undergraduate education worked in intensive care for at least one year, actively continued their profession (no annual leave, report, etc.), and were willing and voluntary to participate in the study were included in the study. Nurses who had a palliative care nursing certificate, had received training on end-of-life care by participating in a training program such as ELNEC, and had not participated in the training program of the study for more than two sessions were not included in the study.

At the beginning of the research, the pre-test forms/scales "Nurse Information Form", "End-of-Life Care Knowledge Test" and "Intensive Care Nurses' Attitudes and Behaviors Towards End-of-Life Care Scale" were administered to all nurses. After the pre-test application, the nurses were randomly included in the training and control groups. A randomization list generated by a computer-based random number sequence was used to determine which group the intensive care nurses would be in.

* The "End-of-Life Care Education Program in Intensive Care" prepared by the researchers in line with the End-of-Life Nursing Education-Intensive Care program was applied to the intensive care nurses in the training group. The training program was implemented online for 45-60 minutes one day a week for 4 weeks. The same forms/scales were repeated 4 weeks after the training.
* Intensive care nurses in the control group did not receive any intervention during the study. Similar to the training group, the same forms/scales were repeated 4 weeks after the training. After the study is completed, the same training program will be applied to the nurses in the control group.

DETAILED DESCRIPTION:
End-of-life care is defined as a support and care program that requires the use of psychosocial skills and techniques to meet the expectations and needs of the patient and his/her family in cases where treatment is no longer possible and to enable the patient and his/her family to live as comfortably as possible in this final period. According to World Health Organization data, more than 30 million individuals have died due to a disease requiring end-of-life care and approximately 20 million of them need intensive care. It is observed that nurses do not have sufficient knowledge and skills in clinical practice due to the lack of importance given to end-of-life care in the nursing education curriculum. In recent studies, it is a remarkable result for intensive care nurses that intensive care nurses cannot define end-of-life care and that their knowledge about end-of-life care is not at the desired level. These results in the literature reveal the importance of end-of-life care education for intensive care nurses. It has been reported that the end-of-life care provided by intensive care nurses to patients and their relatives is affected by nurses' attitudes and behaviors towards end-of-life care as well as their level of knowledge. In addition, examining the attitudes and behaviors of intensive care nurses about providing end-of-life care will guide both the awareness of the problems experienced by nurses and the planning of effective care services. In this context, it will be possible for intensive care nurses to provide holistic and holistic care to the patient and his/her family at the end of life, to meet the psycho-social needs of the patient, to have sufficient knowledge about end-of-life care and to exhibit positive attitudes and behaviors. This study was designed as a randomized controlled trial to evaluate the effect of end-of-life care awareness training to be given to intensive care nurses on their knowledge levels, attitudes, and behaviors.

The sample of the study consisted of intensive care nurses working in the tertiary intensive care units of the University of Health Sciences Van Training and Research Hospital. Sampling calculation was done with G Power 3.1.9.7 package program. The number of nurses included in the study was calculated as a minimum of 34 nurses for each group with 80% power and 5% type 1 error, taking the study of Ghaemizade et al. (2022) as an example. However, in order to secure the sample number and to keep the power value high, the sample number was increased and a total of 76 nurses, including 38 nurses in each group, were included in the sample.

Randomization Method: After obtaining the permission of the ethics committee, patients who meet the inclusion criteria in the study and who have received written informed consent to participate in the study will be divided into two groups in equal numbers with the computer-based randomization method.

Statistical analyses were performed using the SPSS-22 package program. Kolmogorov-Smirnov test, skewness, and kurtosis values were used to test whether the data were normally distributed. Number, percentage, mean, standard deviation, median, and minimum-maximum values were used in descriptive statistics. Independent samples t-tests and chi-square tests were used to compare the demographic characteristics of the two groups. Independent samples t-test was used to compare the mean scores of the dependent variables (end-of-life care knowledge test, attitude, and behavior levels) of the two groups. The t-test for dependent samples and the ANOVA test were used to compare the mean scores of the dependent variables of each group at baseline and 4 weeks (±3 days) after the training (within-group differences). Following the analysis of variance, the "Tukey test" was used to determine different groups. Pearson correlation coefficients were calculated to determine the relationships between continuous measurements. The statistical significance level was taken as 5% in the calculations.

ELIGIBILITY:
Inclusion Criteria:

* Completion of undergraduate education,
* Working in intensive care for at least one year,
* Actively continuing his/her profession (no annual leave, report, etc.)
* Willingness and voluntariness to participate in the research

Exclusion Criteria:

* To have a palliative care nursing certificate,
* Having received training on end-of-life care by participating in a training program such as ELNEC etc,
* Not having attended more than two sessions in the training program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
The End-of-Life Care Knowledge Test | It was used at baseline and 4 weeks (±3 days) after the training program.
  It was prepared by the researcher to evaluate the knowledge levels of intensive care nurses in accordance with the content of the "End-of-Life Care Awareness Training Program".This test consists of 25 questions. The answers have 5 options and there is one correct answer for each question. Each correct answer is scored as 1 (one) point and each incorrect answer is scored as 0 (zero) points. The increase in the number of correct answers to the questions indicates an increase in the level of knowledge.
Attitudes and Behaviors of Intensive Care Nurses Towards End-of-Life Care Scale | It was used at baseline and 4 weeks (±3 days) after the training program.
  It evaluates attitudes towards end-of-life care with 10 questions and behaviors with 6 questions. An increase in the scale score indicates that nurses exhibit positive attitudes and behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Institute of Graduate Studies in Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No